CLINICAL TRIAL: NCT01461421
Title: Acceptance Based Behavioral Intervention for Weight Loss: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Rena R. Wing, Director Weight Control & Diabetes Research Center, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DK087704-01A1 (NIH)
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: Obesity; Primary Care; Behavior Modification
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Behavioral Treatment (Active Comparator): Nutrition education, behavioral weight loss techniques, and standard cognitive strategies for dealing with stress and emotions. Six months weekly, 3 months bi-weekly, 3 months monthly.
  Interventions: Behavioral: Nutrition Education; Behavioral: Behavioral Weight Loss Strategies; Behavioral: Standard Cognitive Techniques
- Acceptance Based Behavioral Intervention (Experimental): Nutrition education, behavioral weight loss techniques, and acceptance based strategies for dealing with stress and emotions. Six months weekly, 3 months bi-weekly, 3 months monthly.
  Interventions: Behavioral: Nutrition Education; Behavioral: Behavioral Weight Loss Strategies; Behavioral: Acceptance Based Techniques

INTERVENTIONS:
Behavioral: Nutrition Education — Participants are taught about energy balance, caloric intake, the nutrition content of foods, and diet.
Behavioral: Behavioral Weight Loss Strategies — Participants are taught self-monitoring and goal setting techniques.
Behavioral: Standard Cognitive Techniques — Participants are taught how to modify, get rid of, or distract from thoughts and also how to regulate emotions.
  Arms: Standard Behavioral Treatment
Behavioral: Acceptance Based Techniques — Participants are taught how to accept and change their perception of their thoughts and emotions.
  Arms: Acceptance Based Behavioral Intervention

SUMMARY:
The proposed project is testing two behavioral interventions designed to improve long-term weight loss among participants who struggle with eating in response to stress or emotional experiences. Group treatment lasts for 1 year, with assessments lasting 2 years. Participants must live in the greater Providence, Rhode Island area in order to be eligible.

DETAILED DESCRIPTION:
Obesity is a major health problem and behavioral weight control programs are the treatment of choice for mild and moderate obesity. However, there is marked variability among participants in the weight losses achieved in these programs and the maximum weight losses are typically achieved at month 6, followed by weight regain. Thus innovative approaches are needed to improve longer-term treatment outcomes.

Currently, the same behavioral treatment program is offered to all participants, with no tailoring to meet the needs of specific subgroups. One subgroup that may need a specialized approach are those who report high levels of internal disinhibition, i.e. eating in response to negative thoughts or emotions. Over 50% of individuals entering behavioral weight loss programs report high levels of internal disinhibition on the Eating Inventory (EI), this subgroup is distinct from those with binge eating disorder, and most importantly, these individuals lose significantly less weight than other participants during weight loss treatment [particularly at 18 months]. Thus efforts are needed to develop more effective treatments for this subgroup. The proposed research is significant because it may help move the field from a "one size fits all" approach, to the development of interventions for specific subgroups of the population.

The investigators hypothesize that individuals who report problems with internal disinhibition may achieve better weight losses in an enhanced behavioral weight loss program that focuses on acceptance-based strategies. Whereas standard behavioral treatments teach patients to control their negative thoughts with techniques such as cognitive restructuring and distraction, acceptance based strategies teach patients to experience thoughts and feelings as they are, without attempting to control them and to continue to pursue their behavioral goals despite experiencing negative thoughts and feelings. Acceptance-based strategies have been shown to be helpful for a number of behavioral problems including weight loss and maintenance, however are yet untested in large trials.

The current study is a randomized controlled trial comparing standard behavioral weight loss treatment with a program which incorporates acceptance based strategies in the treatment of overweight/obese individuals with problems with internal disinhibition. A total of 160 participants will be randomly assigned to a standard behavioral weight loss treatment program (SBT) or to an innovative approach that combines standard behavioral weight loss with acceptance based strategies (referred to hereafter as "Acceptance Based Behavioral Intervention" or ABBI). Both groups will meet weekly for 6 months, biweekly for 3 months and then monthly for 3 months. Assessments will be conducted at baseline and 6 month intervals for 24 months total, with measures of weight, acceptance of negative emotions, distress tolerance, and adherence to the weight loss program.

The primary hypothesis is that participants in the ABBI program will achieve greater changes in weight (in the form of weight reductions) at 6, 12, 18, and 24 months when compared to baseline weight than participants in SBT. Secondary hypotheses are that participants in ABBI will experience greater improvements in acceptance of weight related negative thoughts and emotions and distress tolerance and better treatment adherence than participants in SBT.

ELIGIBILITY:
Inclusion Criteria:

* Must live in the greater Providence, RI area and be able to attend treatment sessions on site for 1 year
* BMI between 30-50
* Age between 18-70
* meets clinical cutoff on Internal Disinhibition sub-scale of the Eating Inventory

Exclusion Criteria:

* report a heart condition, chest pain during periods of activity or rest, or loss of consciousness
* physically unable to exercise
* are currently pregnant or plan to become pregnant in the next 24 months
* are planning to move outside the state within the next 24 months
* Cancer diagnoses in the past 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weight | 6, 12, 18, and 24 months
  Amount of weight lost (kg) from initial body weight at study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Rena R. Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Lillis J, Niemeier HM, Ross KM, Thomas JG, Leahey T, Unick J, Kendra KE, Wing RR. Weight loss intervention for individuals with high internal disinhibition: design of the Acceptance Based Behavioral Intervention (ABBI) randomized controlled trial. BMC Psychol. 2015 May 28;3(1):17. doi: 10.1186/s40359-015-0075-2. eCollection 2015. PMID 26019869